CLINICAL TRIAL: NCT04980404
Title: A Phase Ib Study of Oral Decitabine/Cedazuridine as Maintenance Therapy Following Allogeneic Hematopoietic Cell Transplantation for Patients With Myeloid Neoplasms
Brief Title: Inqovi Maintenance Therapy in Myeloid Neoplasms
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Principal Investigator, Zachariah Michael DeFilipp, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-214
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Stem Cell Leukemia
Keywords: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Stem Cell Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute | interventions — decitabine and cedazuridine drug combination; Decitabine; cedazuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Inqovi (Experimental): Study will follow a standard '3+3' dose escalation design:
  * Initial group of 3 participants will receive Inqovi (decitabine/cedazuridine) on days 1-3 of a 42 day cycle/dose-limiting toxicity (DLT) period.
  * Additional enrollment, dosage and study cyles will be determined by number of dose-limiting toxicity (DLT) that occur in initial group
  Interventions: Drug: Inqovi
- Recommended Phase 2 Dose Expansion (RP2S) Inqovi (Experimental): Once the Recommended Phase 2 Dose Expansion (RP2S) is established, 10 additional participants will be enrolled and receive Inqovi (decitabine/cedazuridine) on days 1-3 of a 28 day study cycle.
  Interventions: Drug: Inqovi

INTERVENTIONS:
Drug: Inqovi — Tablet combination of drugs decitabine and cedazuridine, given orally.
  Other Names: decitabine; cedazuridine

SUMMARY:
This research is being done to see if the drug Inqov is effective in reducing the chance of myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) relapsing after standard of care stem cell transplant.

* This research study involves the study drug Inqovi, which is a combination of the drugs decitabine and cedazuridine.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label, phase Ib study of oral Inqov-decitabine/cedazuridine, given as maintenance therapy following allogeneic hematopoietic cell transplantation for patients with myeloid neoplasms

The U.S. Food and Drug Administration (FDA) has approved Inqovi for myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) relapse but it has not been investigated in the post-transplant setting.

Inqovi is made up of the two study drugs decitabine and cedazuridine. Decitabine is believed to work by stopping cancer cells from growing and spreading. Cedazuridine is believed to work by slowing down how quickly the body breaks down decitabine, which normally breaks down too quickly to be effective.

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

As the study is looking for the highest dose of Inqovi that can be administered safely without severe or unmanageable side effects not everyone will receive the same dose of the study drug. Dosage will depend on the number of participants who have been enrolled in the study before and how well they have tolerated their doses.

Participants will receive study treatment for up to 12 months and will be followed for up to 24 months after starting the study drug.

It is expected that about 22 people will take part in this research study.

Taiho Oncology, Inc., a pharmaceutical company, is supporting this research study by providing funding for the study, including the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML).

  * Subjects should have less than 5% myeloblasts on a bone marrow biopsy within 42 days prior to the start of conditioning.
* Age ≥ 18
* Will undergo first allogeneic hematopoietic stem cell transplantation (HSCT) for their malignancy.
* Transplantation will be performed with the use of reduced intensity conditioning (RIC).
* HSCT Donor will be one of the following:

  * 5/6 or 6/6 (HLA-A, B, DR) matched related donor
  * 7/8 or 8/8 (HLA-A, B, DR, C) matched unrelated donor. Matching in the unrelated setting must be at the allele level.
  * Haploidentical related donor, defined as ≥ 3/6 (HLA-A, B, DR) matched
  * ≥ 4/6 (HLA-A, B, DR) umbilical cord blood (UCB). Matching in the UCB setting is at the antigen level. Recipients may receive either one or two UCB units. In the case of 2 UCB units, both units must have been at least 4/6 matched with the recipient.
* ECOG performance status 0-2.
* Participants must have normal organ and function as defined below:

  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
  * Total bilirubin < 1.5 x ULN (with the exception of subjects with a history of Gilbert's syndrome)
  * Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)
* LVEF must be equal to or greater than 50%, as measured by MUGA scan or echocardiogram
* Female patients of childbearing potential must have a negative pregnancy test, as measured by serum or urine testing
* The effects of decitabine/cedazuridine on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during the entire study treatment period and through 6 months after the last dose of treatment
* Ability to understand and the willingness to sign a written informed consent document.

Eligibility Criteria Prior to Treatment (Post HCT)

* Maintenance therapy may begin at any time between day 30 and day 120 following hematopoietic cell transplantation. Participants must meet the following criteria to be eligible to treatment on this study:

  * Chimerism studies reveal that ≥ 70% of blood or bone marrow cells, or of the CD33 expressing fraction, are of donor origin.
  * There is no acute graft versus host disease (GVHD), requiring an escalation of corticosteroid dose or addition of other agent in the 4 weeks prior to Cycle 1 Day 1.
  * There is no morphological evidence of relapsed/recurrent/residual disease (as assessed by post HCT bone marrow biopsy and aspirate).
  * There is no systemic infection requiring IV antibiotic or antifungal or antiviral therapy within 7 days of starting decitabine/cedazuridine
  * ANC ≥ 1000/µL
  * Platelets ≥ 50,000/µL
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
  * Total bilirubin < 1.5 x ULN (with the exception of subjects with a history of Gilbert's syndrome)
  * Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplants.
* History of other malignancy(ies) unless

  * the participant has been disease-free for at least 12 months and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Known diagnosis of active hepatitis B or hepatitis C
* Current or history of congestive heart failure New York Heart Association (NHYA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 50%, as measured by MUGA scan or echocardiogram)
* Current or history of ventricular or life-threatening arrhythmias or diagnosis of long-QT syndrome
* Systemic uncontrolled infection
* Known dysphagia, short-gut syndrome, gastroparesis, or other condition(s) that limits the ingestion or gastrointestinal absorption of drugs administered orally
* Uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg)
* QTc interval (i.e., Friderica's correction [QTcF]) ≥ 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Schedule Dose | 42 Days
  Identify the recommended phase II schedule of oral decitabine/cedazuridine through standard 3+3 Dose escalation model.

SECONDARY OUTCOMES:
Median number of days of Inqovi tolerated | Up to 2 years
  Median number of day of Inqovi tolerated tabulated and reported descriptively.
Cumulative incidence of acute GVHD | Up to 2 years
  Cumulative incidence of acute GVHD tabulated and reported descriptively.
Cumulative incidence of significant chronic GVHD | Up to 2 years
  Cumulative incidence of significant chronic GVHD tabulated and reported descriptively.
Overall survival Rate | The time from first dose of study drug to the date of death due to any cause up to 2 years
  Assessed using Kaplan-Meier
Relapse-free survival Rate | The time from first dose of study drug to the earlier of relapse or death due to any cause up to 2 years
  Assessed using Kaplan-Meier
Proportion of subjects who successfully screen for study prior to transplantation but who do not reach the maintenance phase due to transplant related morbidity or mortality. | Up to 2 years
  Proportion of subjects who successfully screen for study prior to transplantation but who do not reach the maintenance phase due to transplant related morbidity or mortality tabulated and reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation